CLINICAL TRIAL: NCT05664646
Title: Autonomic Effects of Transcutaneous Spinal Cord Stimulation in Veterans With SCI
Brief Title: Autonomic Effects of Stimulation in SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: B4373-P; 1I21RX004373-01A1 (NIH)
Record Dates: First submitted 2022-12-15; First posted 2022-12-27 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injury
Keywords: Orthostatic Hypotension; Exercise; Hypotension; Body Core Temperature; Blood Pressure
MeSH Terms: conditions — Spinal Cord Injuries; Hypotension, Orthostatic; Motor Activity; Hypotension | interventions — Transcutaneous Electric Nerve Stimulation; Exercise Test

STUDY DESIGN:
Intervention Model Description: During the study 1 visits, the participants will complete an arm ergometry exercise with the optimal stimulation parameters and without (sham). During study 2 visits, the participants' body core temperature will be measured about being exposed to a cool environment with stimulation and without (sham).
Who Masked: Participant
Masking Description: During both Study 1 and Study 2, the participants will be blinded to the order of completing the study with and without stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Without stimulation (Sham Comparator): For study 1, exercise power output and heart rate recovery will be measured after arm ergometry without stimulation. For study 2, body core temperature and thermal comfort will be reported without stimulation.
  Interventions: Other: Arm Ergometry; Other: Cool Environment
- With stimulation (Active Comparator): For study 1, exercise power output and heart rate recovery will be measured after arm ergometry with stimulation. For study 2, body core temperature and thermal comfort will be reported with stimulation.
  Interventions: Device: DS8R; Other: Arm Ergometry; Other: Cool Environment

INTERVENTIONS:
Device: DS8R — transcutaneous stimulation of the spinal cord.
  Other Names: Transcutaneous Stimulation
  Arms: With stimulation
Other: Arm Ergometry — Study 1 will use the arm ergometry as a form of exercise.
  Other Names: Arm cycling
Other: Cool Environment — Study 2 will be completed in a cool environment setting.

SUMMARY:
This study aims to determine the effects of transcutaneous spinal cord stimulation to increase blood pressure and use that device to increase power output and heart rate recovery during arm cycle ergometry. In addition, the investigators will see if the stimulation helps regulate body temperature when in a cool environment.

DETAILED DESCRIPTION:
This study aims to determine the effects of transcutaneous spinal cord stimulation to increase blood pressure and use that device to increase exercise power output and heart rate recovery during arm cycle ergometry. In addition, the investigators will see if the stimulation helps regulate body temperature when in a cool environment. Study 1 (arm cycle ergometry) will consist of 2 visits that will be between 2-3 hours in duration, separated by no less than 3 days, and will consist of putting the electrode at the optimal spot on the spine and completing a submaximal arm ergometry exercise and the other visit will be a sham visit. Study 2 (cool environment) will consist of 2 visits that will be between 3-4 hours in duration, separated by no less than 3 days, and will consist of assessing core temperature when in a cool environment with the stimulator on and off.

ELIGIBILITY:
Inclusion Criteria:

* injury more than 1 year ago, non-ambulatory
* level of lesion C3-T6, AIS A, B, or C
* stable prescription medication regimen for at least 30 days
* must be able to commit to study requirements of 7 visits within a 60-day period

Exclusion Criteria:

* extensive history of seizures
* ventilator dependence or patent tracheostomy site
* history of neurologic disorder other than SCI
* history of moderate or severe head trauma
* contraindications to spine stimulation
* significant cardiovascular disease
* active psychological disorder
* recent history (within 3 months) of substance abuse
* open skin lesions over spine at levels targeted for stimulation (L1/L2) and pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Power Output | through study completion, up to 2 years
  Determine if TSCS increases power output (watts) compared to no stimulation.
Heart Rate Recovery Time | through study completion, up to 2 years
  Determine if TSCS shortens the amount of time for HR recovery (return to baseline) compared to no stimulation.
Total Distance Achieved | through study completion, up to 2 years
  Determine if TSCS increases total distance (miles) achieved during arm ergometry compared to no stimulation.
Body Core Temperature | through study completion, up to 2 years
  Determine if TSCS helps maintain body core temperature in a cool environment compared to no stimulation.

SECONDARY OUTCOMES:
Subjective Reporting on Thermal Comfort and Thermal Sensation | through study completion, up to 2 years
  To determine if TSCS helps improve subjective reporting on thermal comfort and thermal sensation compared to no stimulation.
Exercise Endurance Time | through study completion, up to 2 years
  Determine if TSCS increases exercise endurance time compared to no stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Wecht, EdD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No